CLINICAL TRIAL: NCT04487704
Title: A Real World Study of Treatment Regimens Containing Camrelizumab in Patients With Advanced Liver Cancer
Brief Title: Camrelizumab Utilization on Patients With Advanced Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJYFY-KRLZ-HCC-1
Record Dates: First submitted 2020-05-27; First posted 2020-07-27 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: RWS; Advanced Liver Cancer; PD-1
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Camrelizumab in the treatment of liver cancer (Other): Camrelizumab intravenous infusion (no need for prophylactic administration), no less than 30 min
  Interventions: Other: camrelizumab

INTERVENTIONS:
Other: camrelizumab — camrelizumab 200 mg, intravenous infusion (no need for prophylactic administration), no less than 30 min ，No more than 60 min, one cycle every 2 weeks (14 days) or one cycle every 3 weeks (21 days). Try to complete the administration before the ECG

SUMMARY:
To observe and evaluate the safety and efficacy of camrelizumab in advanced liver cancer

DETAILED DESCRIPTION:
camrelizumab ， a humanized monoclonal antibody against PD-1, has been shown to block the binding of PD-1 to PD-L1, thereby inhibiting the immune escape of tumor cells. It has a high affinity for PD-1 (KD = 3.31 nmol/L), a high acceptor proportion (85% at 200 mg) of circulating T lymphocytes, and binds to epitopes different from Nivolumab and pembrolizumab，Phase 1 clinical trials have shown that camrelizumab is well tolerated and has antitumor activity in patients with advanced solid tumors.camrelizumab has been approved for indication for advanced hepatocellular carcinoma The main objective of this study was to observe and evaluate the safety and efficacy of treatment regiments containing Camrelizumab in advanced liver cancer。 The subjects included people over 18 years old， For men and women with advanced liver cancer confirmed by histopathology or cytology;

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more;
* For both men and women;
* Patients with advanced liver cancer confirmed by histopathology or cytology; .Volunteer to join the study, sign the informed consent, good compliance, and cooperate with the follow-up.

Exclusion Criteria:

* A known allergy to the study drug or any of its excipients; Or had a severe allergic reaction to other monoclonal antibodies;
* Patients who are ready for or have previously received an organ or allogeneic bone marrow transplant;
* Pregnant or lactating women;
* According to the judgment of the researcher, the patients should not be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Assess Safety as defined by the NCI CTCAE v5.0 | From patients participate in the clinical study to 90 days after the end of treatment
  Adverse events as graded by CTCAE v5.0

SECONDARY OUTCOMES:
overall survival | 5 years
  1-year, 3-year, 5-year survival

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lyu, MD,phD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China